CLINICAL TRIAL: NCT04705350
Title: A Randomized, Participant-Blind, Investigator-Blind, Placebo-Controlled Study Evaluating Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Intravenous Doses of Zampilimab in Healthy Participants
Brief Title: A Study to Test Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Intravenous Doses of Zampilimab in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UP0105; 2020-004411-26 (EudraCT Number)
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Healthy Study Participants
Keywords: Healthy study participants; UCB7858; zampilimab; Phase 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a participant- and Investigator-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zampilimab Cohorts (Experimental): Participants will be randomized to receive predefined single doses of zampilimab.
  Interventions: Drug: Zampilimab
- Placebo (Placebo Comparator): Participants randomized to this arm will receive matching Placebo to maintain the blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zampilimab — Participants will receive a single intravenous dose of zampilimab at a pre-specified time point.
  Other Names: UCB7858
  Arms: Zampilimab Cohorts
Drug: Placebo — Participants will receive matching placebo at a pre-specified time point to maintain the blinding.
  Other Names: PBO
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics (PK) of zampilimab in healthy study participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the Informed Consent Form (ICF)
* Study participant must be considered reliable and capable of adhering to the protocol, according to the judgment of the Investigator, and is able to communicate satisfactorily with the Investigator and comply with all clinical study requirements
* Study participant has adequate peripheral venous access
* Study participant has clinical laboratory test results within the reference ranges of the testing laboratory. Study participants with test results that are outside the specified ranges and that are deemed as clinically nonsignificant will be allowed at the discretion of the Investigator
* Study participant is of normal weight as determined by a body mass index between 18 and 32 kg/m^2, inclusive, with a body weight of at least 50 kg (male) or 45 kg (female) and no greater than 100 kg
* Study participants may be male or female
* Male participants must agree to use contraception during treatment period and for 5 months; female participants of childbearing potential must be not pregnant or breastfeeding and agree to use contraception during the treatment period and for 5 months

Exclusion Criteria:

* Study participant has any medical (acute or chronic) or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the IMP; or interfering with the interpretation of data
* Study participant has a known hypersensitivity to any components of the investigational medicinal product (IMP) as stated in this protocol or participant has a history of moderate to severe allergic reaction to medication(s), including biologics
* Study participant has any clinically relevant abnormal findings in physical examination, laboratory tests, vital signs, or electrocardiogram (ECG), which, in the opinion of the Investigator, may place the participant at risk because of participation in the study
* Study participant has had major surgery (including joint surgery) within 6 months prior to the Screening Period, or has planned surgery within 6 months after IMP
* Study participant has current diagnosis or history of wound healing complications
* Study participant has a history of alcohol and/or drug abuse up to 6 months before the Screening Period
* Study participant has active neoplastic disease or history of neoplastic disease within 5 years of the Screening Period
* Study participant has an active infection during the Screening Period
* Study participant has clinical signs and symptoms consistent with coronavirus disease (COVID-19) or had a positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test result within the last 4 weeks prior to the Screening Period or on admission
* Study participant has had a severe course of COVID-19 that required hospitalization
* Study participant has received any prescription or nonprescription medicines, including over the counter (OTC) remedies or herbal and dietary supplements, within 14 days or 5 half-lives of the respective drug, whichever is longer, other than the occasional use of analgesics, such as paracetamol (acetaminophen) or ibuprofen, oral contraceptives, or inhaled corticosteroids for seasonal rhinitis
* Study participant has received treatment with biologic agents (such as monoclonal antibodies (mAbs) including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing
* Study participant has received a vaccination within 8 weeks prior to Day 1; or intends to have a vaccination during the course of the study
* Study participant has participated in another study of a IMP (and/or an investigational device) within the previous 3 months or 5 half-lives prior to the Screening Period, whichever is longer, or is currently participating in another study of a IMP (and/or an investigational device)
* Study participant has positive serology test for hepatitis B surface antigen, hepatitis B core antibodies (both immunoglobulin G (IgG) and IgM), hepatitis C virus antibodies, or antibodies to human immunodeficiency virus type 1 and/or type 2 during the Screening Period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Incidents of treatment-emergent adverse events (TEAEs) through the Safety Follow-up (SFU) Visit | From Day 1 (Start of Treatment Period) to the end of Safety Follow-up (up to 120 days)
  A treatment-emergent adverse event (TEAE) is defined as any event not present prior to the administration of investigational medicinal product (IMP) or any unresolved event already present before administration of IMP that worsens in intensity following exposure to the treatment.
Maximum intensity of treatment-emergent adverse events (TEAEs) through the Safety Follow-up (SFU) Visit | From Day 1 (Start of Treatment Period) to the end of Safety Follow-up (up to 120 days)
  Maximum intensity across all incidents of each TEAE for each study participant

SECONDARY OUTCOMES:
Maximum zampilimab serum concentration (Cmax) | From Day 1 (Start of Treatment Period) to the end of Safety Follow-up (up to 120 days)
  Cmax: Maximum observed zampilimab serum concentration
Time to maximum zampilimab serum concentration (tmax) | From Day 1 (Start of Treatment Period) to the end of Safety Follow-up (up to 120 days)
  tmax: Time to maximum observed zampilimab serum concentration
Area under the zampilimab serum concentration-time curve from time zero to last quantifiable concentration (AUC0-t) | From Day 1 (Start of Treatment Period) at predefined time points to the last quantifiable concentration (up to 120 days)
  AUC0-t: Area under the zampilimab serum concentration-time curve from time zero (Day 1) to the last quantifiable concentration
Area under the zampilimab serum concentration-time curve from time zero to infinity (AUC) | Day 1 (Start of Treatment Period) at predefined time points (up to 120 days)
  AUC: Area under the zampilimab serum concentration-time curve from time 0 (Day 1) to infinity
Clearance (CL) of zampilimab in serum | From Day 1 (Start of Treatment Period) to the end of Safety Follow-up (up to 120 days)
  CL: volume of serum that is cleared from zampilimab per unit of time
Apparent volume of distribution during terminal phase (Vz) of zampilimab | From Day 1 (Start of Treatment Period) to the end of Safety Follow-up (up to 120 days)
  Vz: apparent volume of distribution during terminal phase
Apparent terminal half-life (t1/2) of zampilimab | From Day 1 (Start of Treatment Period) to the end of Safety Follow-up (up to 120 days)
  t1/2: terminal zampilimab serum half-life

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Principal Investigator — 001 844 599 2273 (UCB)
Locations (1):
- Up0105 001, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.